CLINICAL TRIAL: NCT00943657
Title: An Open-Label Phase 3 Study to Assess the Immunogenicity and Safety of a Vero Cell-Derived Trivalent Seasonal Influenza Vaccine, Strain Composition 2009/2010, in an Adult and Elderly Population
Brief Title: Yearly Strain Variation Study, 2009/2010
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alachua Government Services, Inc. (Industry)
Responsible Party: Gerald Aichinger, MD; Study Medical Director, Baxter Healthcare Corporation
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 720901
Record Dates: First submitted 2009-07-21; First posted 2009-07-22 (Estimated); Last update posted 2015-10-09 (Estimated); Status verified 2009-10

CONDITIONS: Influenza; Seasonal Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: Preflucel [Trivalent seasonal influenza vaccine (split virus, Vero cell-derived)] — Single intramuscular injection of vaccine
  Other Names: Preflucel

SUMMARY:
The purpose of this study is to verify the immunogenicity and tolerance of a trivalent seasonal influenza vaccine with strain composition according to World Heath Organization/European Union (WHO/EU) recommendation for the 2009/2010 season for yearly licensing application.

ELIGIBILITY:
Inclusion Criteria:

* Subject is 18 to 59 years of age , inclusive, at the time of screening (for subjects in age stratum A only)
* Subject is 60 years of age or older , inclusive, at the time of screening (for subjects in age stratum B only)
* Subject has given written informed consent prior to study entry
* Subject is generally healthy , as determined by the investigator's clinical judgment through collection of medical history and performance of a physical examination, such that the investigator would not hesitate to provide routine influenza immunization to the subject in the course of routine medical practice
* Subject agrees to keep a daily record of symptoms for the duration of the study
* If female of childbearing potential, subject presents with a negative urine pregnancy test, and agrees to employ adequate birth control measures for the duration of the study
* Subject is willing and able to comply with the requirements of the protocol

Exclusion Criteria:

* Subject has a history of severe allergic reaction or anaphylaxis
* Subject has an oral temperature of >= 37.5°C on the day of vaccination in this study
* Subject has a rash or dermatologic condition or tattoos, which may interfere with injection site reaction rating
* Subject has received a live vaccine within 4 weeks or an inactivated or subunit vaccine within 2 weeks of study entry
* Subject has received a seasonal influenza vaccine within 6 months of study entry
* Subject currently has or had a history of a significant neurological, cardiovascular, pulmonary (including asthma), hepatic, metabolic, rheumatic, autoimmune, hematological or renal disorder
* Subject has any inherited or acquired immunodeficiency
* Subject has a disease or is currently undergoing a form of treatment or was undergoing a form of treatment within 30 days prior to study entry that can be expected to influence immune response. Such treatment includes, but is not limited to, systemic or high dose inhaled (>800 µg/day of beclomethasone dipropionate or equivalent) corticosteroids, radiation treatment or other immunosuppressive or cytotoxic drugs.
* Subject has a functional or surgical asplenia
* Subject has a known or suspected problem with alcohol or drug abuse
* Subject is a member of the team conducting this study or is in a dependent relationship with one of the study team members. Dependent relationships include close relatives (ie, children, partner/spouse, siblings, parents) as well as employees of the investigator or site personnel conducting the study
* If female, subject is pregnant or lactating at the time of study enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2009-06; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Number of subjects demonstrating seroconversion to each of the three antigens contained in the vaccine 21 days after vaccination | 21 days

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Department of Clinical Pharmacology, Vienna, Austria